CLINICAL TRIAL: NCT01291459
Title: Phase II Pilot Study of Simplification to Maraviroc - Raltegravir Dual Therapy After 6 Months of Maraviroc - Raltegravir - Tenofovir - Emtricitabine Quadruple Therapy in ARV Treatment-naive, HIV-1-infected Patients With CCR5- Virus
Brief Title: Pilot Study of Maraviroc/Raltegravir for Naive HIV-1 Patients
Acronym: NNNB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association Pour la Recherche en Infectiologie (Other)
Responsible Party: Principal Investigator, Dr Laurent COTTE, MD, Association Pour la Recherche en Infectiologie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/HD/01
Record Dates: First submitted 2011-01-26; First posted 2011-02-08 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: HIV
Keywords: HIV; naive patients; maraviroc; raltegravir
MeSH Terms: interventions — Raltegravir Potassium; Maraviroc; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Maraviroc/raltegravir/emtricitabine/tenofovir 24 weeks followed by Maraviroc/Raltegravir 24 weeks
  Interventions: Drug: MVC/RAL/FTC/TDF followed by Maraviroc/Raltegravir

INTERVENTIONS:
Drug: MVC/RAL/FTC/TDF followed by Maraviroc/Raltegravir — MVC/RAL/FTC/TDF 24W followed by MVC/RAL until W48.
  Other Names: Maraviroc; Raltegravir; Emtricitabine; Tenofovir

SUMMARY:
Background and Rationale

Raltegravir and Maraviroc, the first in class of 2 new families of antiretroviral drugs have demonstrated a high potency in treatment experienced and naive patients. Both drugs appeared well tolerated with low metabolic toxicity. No data are currently available concerning the combination of these 2 drugs.

Hypothesis

Maraviroc + Raltegravir should be potent enough to maintain virological efficacy in naive patients infected by CCR5 HIV-1 previously treated for 6 months with a Maraviroc-Raltegravir-Tenofovir-Emtricitabine combination.

DETAILED DESCRIPTION:
Objectives:

* To establish the ability of a Maraviroc-Raltegravir combination to maintain HIV-1 viral load < 50 copies/ml at week 48 in naive patients infected by CCR5 HIV-1, following an initial 6 month phase of Maraviroc-Raltegravir-Tenofovir-Emtricitabine combination (Intent to treat and strategy analysis)
* To study CD4 progression from baseline to week 48
* To study the time to virological failure during the simplification phase of the study (from week 24 to week 48)
* To study the proportion of patients with HIV RNA < 50 copies/ml at each time point
* To study the kinetics of viral load decrease from baseline to week 12
* To study the kinetics of proviral DNA decrease from baseline to week 12, 24, 36 and 48
* To study the clinical and biological tolerance of Maraviroc-Raltegravir combination through week 48

Study Design/ Clinical Plan

Pilot, multicenter, national, uncontrolled study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the run-in visit
* HIV-1 infection
* Antiretroviral treatment-naive
* CD4 ≥ 200 /mm3
* HIV- RNA ≥ 1000 copies/ml
* HIV-RNA ≤ 100,000 copies/ml
* Antiretroviral therapy is indicated according to current guidelines
* CCR5-tropic virus according to the Trofile ES® assayGeno2Pheno algorithm using a predefined false positive rate of 20%
* No significant NRTI, NNRTI or PI resistance mutation
* Freely-given, written, informed consent obtained; the patient and investigator have signed the consent form (by the latest on the day of the run-in visit and before performing any examinations required by the trial)
* Patient covered by a French national health insurance scheme

Exclusion Criteria:

* Women of child-bearing potential not using effective contraception (barrier method)
* Pregnant or breast-feeding women
* Patients under the age of 18 years
* Patients deprived of liberty by a judicial or administrative, hospitalized patients without consent, patients admitted to a health or social purposes other than research
* Persons major subject of a measure of legal protection or unable to consent
* Previous antiretroviral therapy (with the exception of post-exposure prophylaxis if HIV serology is negative > 3 months after the last dose of antiretroviral drugs)
* CXCR4-tropic virus, dual/mixed-tropic virus or undetermined tropism on screening
* Presence of significant NRTI, NNRTI or PI resistance mutation(s)
* Infection or co-infection with HIV-2, or group O or N HIV-1
* Acute phase of an opportunistic infection
* Undergoing treatment for tuberculosis
* Undergoing chemotherapy and/or radiotherapy for neoplastic disease
* Decompensated cirrhosis (Child-Pugh class B or C)
* HIV-HBV co-infection. Patients with HIV-HCV co-infection are permitted to participate in the absence of decompensated cirrhosis (Child-Pugh class B or C), of hepatocytolysis > 3 times the upper limit of normal and if treatment for HCV during the ensuing 12 months is not indicated. PAtients with occult HBV are excluded.( positive AcHBc, negative AcHBs, negative AgHBs, positive HBV DNA)
* Co-administration of prohibited treatments (see the SPCs of each product) Laboratory parameters: Haemoglobin < 7g/dl, neutrophil count < 500/mm3, platelet count < 50,000/mm3, creatinine clearance < 50 ml/min, alkaline phosphatase, AST, ALT or bilirubin ≥ 3 times upper limit of normal
* Patient refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
HIV-1 viral load | 48 weeks
  measure of HIV viral load at 48 weeks of treatment for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Laurent COTTE, MD, Principal Investigator
Locations (12):
- France (12):
  - Cannes hosipital, Cannes
  - CHU, Clermont-Ferrand
  - Frejus hospital, Fréjus
  - Edourad Herriot hospital, Lyon
  - Croix Rousse hospital, Lyon
  - Ste MArguerite Hospital, Marseille
  - Conception hospital, Marseille
  - Hotel Dieu hospital, Nantes
  - Hopital l'Archet 1, Nice
  - St Louis Hospital, Paris
  - Pitie Salpetriere Hospital, Paris
  - Nord Hospital, Saint-Etienne